CLINICAL TRIAL: NCT03584581
Title: Effects on Lipid Metabolism of Olive Extracts Rich in Polyphenols
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Ernesto Cortés-Castell, Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI2016/13 nº 77
Record Dates: First submitted 2018-06-27; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Cholesterol; Metabolic Disorder; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive polyphenols (Experimental)
  Interventions: Dietary Supplement: Olive polyphenols
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Olive polyphenols — The amount of polyphenols to be supplied is within the ranges of absolute biosecurity food described by different authors and used in different studies.
  Arms: Olive polyphenols
Dietary Supplement: Control — Placebo
  Arms: Control

SUMMARY:
This study is designed to determine whether a standardized intervention in the health center and based on hygienic dietary measures and physical exercise, supplemented with a polyphenol extract in patients, achieves a greater benefit in the reduction of LDL cholesterol in dyslipidemias in the short term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyslipidemia without the need for pharmacological treatment, but with annual follow-up of their dyslipidemia and with baseline LDL-cholesterol values.
* Patients to whom the annual analysis will be carried out for control of the lipid profile and who agree to postpone it during the month of the health education study.
* Patients who undergo hygienic-dietetic intervention and exercise.
* Patients willing to ingest the nutritional supplement of polyphenols that will be supplied to them.
* Signed the informed consent.

Exclusion Criteria:

* <18 years old.
* High cardiovascular risk.
* With pharmacological treatment.
* With some previous chronic disease.
* With some allergy to the compounds of the product and placebo according to the technical specifications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Cholesterols levels | 1 month
  TC, HDL-C, LDL-C and TG.

SECONDARY OUTCOMES:
BMI (kg/m2) | 1 month
  Weight and height will be combined to report BMI in kg/m^2
Blood pressure | 1 month
  SBP and DBP.
Waist circumference (cm) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital of Elda, Elda, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The data will not be publicly available.

REFERENCES:
- [Background] Tangney CC, Rasmussen HE. Polyphenols, inflammation, and cardiovascular disease. Curr Atheroscler Rep. 2013 May;15(5):324. doi: 10.1007/s11883-013-0324-x. PMID 23512608
- [Background] Bleys J, Miller ER 3rd, Pastor-Barriuso R, Appel LJ, Guallar E. Vitamin-mineral supplementation and the progression of atherosclerosis: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2006 Oct;84(4):880-7; quiz 954-5. doi: 10.1093/ajcn/84.4.880. PMID 17023716
- [Background] Halliwell B, Rafter J, Jenner A. Health promotion by flavonoids, tocopherols, tocotrienols, and other phenols: direct or indirect effects? Antioxidant or not? Am J Clin Nutr. 2005 Jan;81(1 Suppl):268S-276S. doi: 10.1093/ajcn/81.1.268S. PMID 15640490
- [Background] Obied HK, Prenzler PD, Konczak I, Rehman AU, Robards K. Chemistry and bioactivity of olive biophenols in some antioxidant and antiproliferative in vitro bioassays. Chem Res Toxicol. 2009 Jan;22(1):227-34. doi: 10.1021/tx8004168. PMID 19099401
- [Background] Covas MI, Fito M, Lamuela-Raventos RM, Sebastia N, de la Torre-Boronat C, Marrugat J. Virgin olive oil phenolic compounds: binding to human low density lipoprotein (LDL) and effect on LDL oxidation. Int J Clin Pharmacol Res. 2000;20(3-4):49-54. PMID 11314237
- [Background] Veciana Galindo C, Cortes Castell E, Torro Montell L, Sirvent Segura E, Rizo Baeza MM, Gil Guillen V. [Assessment of cytotoxicity and biosafety of polyphenolic extracts from olive pits]. Nutr Hosp. 2014 Jun 1;29(6):1388-93. doi: 10.3305/nh.2014.29.6.7141. Spanish. PMID 24972479
- [Background] Cortes Castell E, Veciana Galindo C, Torro Montell L, Sirvent Segura E, Rizo Baeza MM, Gil Guillen V. [Anti-inflammatory activity of olive seed polyphenolic extract in the THP1-XBLUE-CD14 human monocytes cell line]. Nutr Hosp. 2014 Jul 1;30(1):113-7. doi: 10.3305/nh.2014.30.1.7482. Spanish. PMID 25137269
- [Background] Veciana-Galindo C, Cortes-Castell E, Torro-Montell L, Palazon-Bru A, Sirvent-Segura E, Rizo-Baeza MM, Gil-Guillen VF. Anti-adipogenic activity of an olive seed extract in mouse fibroblasts. Nutr Hosp. 2015 Jun 1;31(6):2747-51. doi: 10.3305/nh.2015.31.6.8997. PMID 26040391
- [Background] Cortes Castell E, Veciana Galindo C, Torro Montell L, Sirvent Segura E, Rizo Baeza MM, Gil Guillen V. [Effect on zebrafish neurodevelopment and neuroprotection of a polyphenolic extract olive seeds]. Nutr Hosp. 2014 Aug 1;30(2):338-42. doi: 10.3305/nh.2014.30.2.7604. Spanish. PMID 25208788
- [Background] Perrinjaquet-Moccetti T, Busjahn A, Schmidlin C, Schmidt A, Bradl B, Aydogan C. Food supplementation with an olive (Olea europaea L.) leaf extract reduces blood pressure in borderline hypertensive monozygotic twins. Phytother Res. 2008 Sep;22(9):1239-42. doi: 10.1002/ptr.2455. PMID 18729245